CLINICAL TRIAL: NCT03184142
Title: Increasing Reporting of Intimidation of Medical Students With Simulation: a Randomised Controlled Trial
Brief Title: Increasing Reporting of Intimidation of Medical Students With Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Érica Patocskai, Surgical Oncologist, Director of surgical Clerkship, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16.422
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Intimidation
Keywords: Intimidation; Simulation; Medical education; Surgical education
MeSH Terms: interventions — Videotape Recording; Control Groups

STUDY DESIGN:
Intervention Model Description: Single-blind randomised controlled trial with two experimental arms and a control arm
Who Masked: Investigator, Outcomes Assessor
Masking Description: Students cannot be masked as an arm undergoes a simulation intervention. The researcher evaluating the outcomes through the questionnaires will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simulation (Experimental): During a suturing class at the simulation center, the students enter a classroom. Although the students are not aware of this, among them is an actor playing the role of a student. One of the two professors is also an actor. As the activity progresses, the professor targets the student played by an actor. The intimidation intensifies until the end. At the end of the activity, there is a debriefing explaining to the students that the bullying professor and the victim were actors.
  Interventions: Behavioral: Simulation
- Video (Experimental): During a suturing class at the simulation center, after 55 minutes of suturing, the students will be exposed to a 15-minute video on workplace and hospital intimidation and how to manage it.
  Interventions: Behavioral: Video
- Control (Placebo Comparator): During a suturing class at the simulation center, the students suture for the entire 70-minute duration of the activity. They are not exposed to intimidation (control group).
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Simulation — Students witness the intimidation of one of their peers (who is an actor) by a professor (also an actor). (see arm description)
  Arms: Simulation
Behavioral: Video — Student watch a 15-minute intimidation video (see arm description).
  Arms: Video
Behavioral: Control group — No intervention. The students suture for 70 minutes
  Arms: Control

SUMMARY:
Intimidation of medical students by health care professionals is a well-documented phenomenon. Raising awareness of what constitutes intimidation is a preferred method for preventing it through increased reporting. Simulation is a novel method of raising awareness of intimidation.

This is a randomised controlled trial comparing the effectiveness of simulation (involving actors), an educational video and no intervention, as adjuncts to group discussion, on students' ability to identify and report intimidation. Medical students from the University of Montreal in Montreal, Canada, will be recruited at the beginning of surgical clerkship. They will complete a standardized and validated pre-intervention questionnaire on their experience with intimidation consisting of multiple choice questions and short answers. They will be randomised to one of the three interventions lasting 70 minutes that will be followed by a 20-minute standardized discussion on intimidation with all students participating together. At the end of their surgical rotation, they will complete a similar post-intervention questionnaire with additional questions pertaining to the reporting of intimidation.

Differences in intimidation reporting after the intervention as well as a before and after comparison of the "Negative Acts Questionnaire" score will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Medical students at the University of Montreal at the beginning of their surgical clerkship rotation.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Comfort in reporting intimidation | 6 weeks after enrollment
  Based on post-intervention questionnaire question.
Perception of intimidation after intervention | 6 weeks after enrollment
  Based on post-intervention Negative Acts Questionnaire (NAQ-R)

SECONDARY OUTCOMES:
Baseline prevalence of intimidation | at enrollment
  Based on pre-intervention Negative Acts Questionnaire (NAQ-R)
Before and after comparison | at enrollment vs 6 weeks post-intervention
  Difference between pre and post-intervention Negative Acts Questionnaire (NAQ-R)
Reasons for not reporting intimidation | at enrollment
  Open-ended question asking why students don't report intimidation
Frequency of intimidation reporting | 6 weeks post-intervention
  Did the students report intimidation during the 6 weeks of their surgical clerkship?

CONTACTS AND LOCATIONS:
Overall Officials: Erica Patocskai, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Faculté de Médecine de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone JP, Charette JH, McPhalen DF, Temple-Oberle C. Under the knife: medical student perceptions of intimidation and mistreatment. J Surg Educ. 2015 Jul-Aug;72(4):749-53. doi: 10.1016/j.jsurg.2015.02.003. PMID 26073477
- [Background] Isaranuwatchai W, Brydges R, Carnahan H, Backstein D, Dubrowski A. Comparing the cost-effectiveness of simulation modalities: a case study of peripheral intravenous catheterization training. Adv Health Sci Educ Theory Pract. 2014 May;19(2):219-32. doi: 10.1007/s10459-013-9464-6. Epub 2013 Jun 1. PMID 23728476
- [Background] Curtis MT, DiazGranados D, Feldman M. Judicious use of simulation technology in continuing medical education. J Contin Educ Health Prof. 2012 Fall;32(4):255-60. doi: 10.1002/chp.21153. PMID 23280528
- [Background] Einarsen S, Helge H, Notelaers G. Measuring exposure to bullying and harassment at work: validity, factor structure & psychometric properties of the negative acts questionnaire-revised. Work Stress 23(1):24-44, 2009.